CLINICAL TRIAL: NCT00790543
Title: Risk Stratification and Identification of Immunogenetic and Microbial Markers of Rapid Disease Progression in Children With Crohn's Disease
Brief Title: Risk Stratification of Rapid Disease Progression in Children With Crohn's Disease
Acronym: RS
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Subra Kugathasan, MD, Professor, Emory University
Other Study IDs: IRB00012206
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At time of enrollment, whole blood for DNA and serum will be collected in all patients. Fresh fecal samples will also be requested. For gene expression analysis, biopsy specimens will be collected during regularly scheduled endoscopies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Children newly diagnosed with Crohn's disease.

SUMMARY:
The purpose of this study for children with a new diagnosis of Crohn's disease is to identify biomarkers found in the blood or stool to help predict which children are at risk of developing complications.

DETAILED DESCRIPTION:
It is estimated that between 15-20% of children with Crohn's disease will develop complications that can require surgery within the first three years of diagnosis. The purpose of this study for children with a new diagnosis of Crohn's disease is to identify biomarkers found in the blood or stool to help predict which children are at risk of developing complications.

A total of 2000 children with newly-diagnosed Crohn's disease will be enrolled within 30 days of diagnosis. Up to 28 medical sites in the United States and Canada will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females younger than 17 years of age (before their 17th birthday). An upper limit of 17 years of age was selected as important inclusion criteria to maximize the number of potential subjects that would be diagnosed and followed by a pediatric gastroenterologist for at least 3 years.
* Confirmed or suspected diagnosis of Crohn's disease based on standardized diagnostic criteria. The enrollment should occur within 30 days of diagnosis.
* Able to provide written informed consent or the ability to obtain written informed consent from the parents or patient's legal guardian in conjunction with youth assent.
* Consented to have specimens tested for genetics and immune responses.
* Access to follow-up data for a minimum of 36 months after diagnosis.
* Final eligibility will be determined by the health professionals conducting this clinical trial.

Exclusion Criteria:

* Infectious colitis.
* Final eligibility will be determined by the health professionals conducting this clinical trial.

Ages: 5 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population will consist of children newly diagnosed with Crohn's disease at primary care clinics.
Sampling Method: Probability Sample
Enrollment: 1813 (Actual)
Dates: Start 2008-11; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Identify demographic, clinical, microbial, genetic, and/or immunologic risk factors influencing the likelihood of rapid development of complicated disease phenotypes manifested as penetrating or stricturing disease and need for surgery. | 3 years

SECONDARY OUTCOMES:
Develop and validate risk stratification by stratifying patients into different levels of risk at diagnosis based on clinical, demographic, host microbial ecology, immune, and genetic determinants. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Subra Kugathasan, MD, Principal Investigator — Emory University
Locations (28):
- United States (25):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Clinic, Jacksonville, Florida
  - Emory-Children's Center - Emory University School of Medicine, Atlanta, Georgia
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Riley Children's Hospital - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Children's Hospital Boston - Harvard Medical School, Boston, Massachusetts
  - Goryeb Children's Hospital - Atlantic Health System, Morristown, New Jersey
  - The Research Foundation of SUNY on behalf of the University at Buffalo, Buffalo, New York
  - Cohens (Schneider) Children's Hospital, New Hyde Park, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Children's Medical Center, Dallas, Texas
  - BCM Texas Children's Hospital - Houston, Houston, Texas
  - Primary Children's Medical Center - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children - Sickkids, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballengee CR, Stidham RW, Liu C, Kim MO, Prince J, Mondal K, Baldassano R, Dubinsky M, Markowitz J, Leleiko N, Hyams J, Denson L, Kugathasan S. Association Between Plasma Level of Collagen Type III Alpha 1 Chain and Development of Strictures in Pediatric Patients With Crohn's Disease. Clin Gastroenterol Hepatol. 2019 Aug;17(9):1799-1806. doi: 10.1016/j.cgh.2018.09.008. Epub 2018 Sep 10. PMID 30213581